CLINICAL TRIAL: NCT04938869
Title: Effect of Continuous Glucose Monitor Application Following Hospital Discharge of Poorly Controlled Patients With Type 2 Diabetes and Active Malignancy
Brief Title: Continuous Glucose Monitor Application After Hospital Discharge for the Improvement of Outcomes in Patients With Poorly Controlled Type 2 Diabetes and Active Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Kathleen Dungan, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-21093; NCI-2021-06008 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-06-17; First posted 2021-06-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (CGM) (Experimental): Prior to hospital discharge, patients receive CGM application and education on how to apply the CGM, and how to use the sensor and its associated smart phone app. Patients also receive basic diabetes mellitus education. After hospital discharge, patients use CGM for up to 28 days.
  Interventions: Other: Educational Intervention; Other: Medical Device Usage and Evaluation; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Receive basic diabetes mellitus education
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Medical Device Usage and Evaluation — Use CGM device and app
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies the effect of a continuous glucose monitor application in improving outcomes in patients with poorly controlled type 2 diabetes and active cancer. Patient satisfaction with type 2 diabetes management influences medication-taking behavior as well as health outcomes. Adding continuous glucose monitor application to diabetes treatment plan after hospital discharge plan may improve patient satisfaction and reduce diabetes distress.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate if addition of continuous glucose monitor (CGM) to diabetes treatment plan following inpatient hospitalization is associated with improved patient satisfaction with DM management in patients with cancer and poorly controlled type 2 diabetes mellitus.

SECONDARY OBJECTIVES:

I. Evaluate feasibility of CGM initiation upon hospital discharge. II. Evaluate effect of CGM on recognition of post-hospitalization hypoglycemia. III. Evaluate patient reported outcome of CGM incorporation into patient diabetes care burden.

IV. Evaluate effect of CGM on depression score before and after CGM use.

OUTLINE:

Prior to hospital discharge, patients receive CGM application and education on how to apply the CGM, and how to use the sensor and its associated smart phone application (app). Patients also receive basic diabetes mellitus education. After hospital discharge, patients use CGM for up to 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Insulin use > 10 units per day
* Hemoglobin A1c > 8.5%
* Smart phone compatible with LibreView App

Exclusion Criteria:

* Type 1 diabetes mellitus (DM)
* Inability to consent
* Pregnancy
* Prisoners
* Discharge to skilled nursing facility

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Change in Diabetes Treatment Satisfaction Questionnaire (DTSQ) survey score | From baseline to 4 weeks post-discharge
  Descriptive statistics will summarize the sample characteristics and distribution of each variable. Change over time in continuous variables will be reported as paired t-test or nonparametric test as appropriate.

SECONDARY OUTCOMES:
Change in DTSQ scores | From baseline to 2 weeks post-discharge
  Descriptive statistics will summarize the sample characteristics and distribution of each variable. Change over time in continuous variables will be reported as paired t-test or nonparametric test as appropriate.
Overall control | Up to 4 weeks post-discharge
  Descriptive statistics will summarize the sample characteristics and distribution of each variable.
Change in various measures of control | From week 1 to week 4
  Descriptive statistics will summarize the sample characteristics and distribution of each variable. Change over time in continuous variables will be reported as paired t-test or nonparametric test as appropriate.
Number of patients with successful data collection | At 2 weeks
  Descriptive statistics will summarize the sample characteristics and distribution of each variable.
Number of patients with successful data collection | At 4 weeks
  Descriptive statistics will summarize the sample characteristics and distribution of each variable.
Change in Patient Health Questionnaire scores | From baseline to 4 weeks post-discharge
  Descriptive statistics will summarize the sample characteristics and distribution of each variable. Change over time in continuous variables will be reported as paired t-test or nonparametric test as appropriate.
Incidence of adverse events | Immediately following inpatient hospitalization
  Will report the safety of continuous glucose monitor application and use. Descriptive statistics will summarize the sample characteristics and distribution of each variable.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Dungan, MD, MPH, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu